CLINICAL TRIAL: NCT05589324
Title: The Effectiveness of Different Angle of 3D Printing Writing Assisitive Device on Feasibility in Patients With Nerve Injury
Brief Title: Effects of 3D Printing Writing Assisitive Device on Feasibility in Patients With Nerve Injury
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Hsinchieh Lee, Principal Investigator, Taipei Medical University Shuang Ho Hospital
Other Study IDs: TMU-JIRB N202206087
Record Dates: First submitted 2022-07-27; First posted 2022-10-21 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Nerve Injury

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3D-printed writing aids group: Thirty subjects were recruited from outpatient rehabilitation of neurologically injured patients with limited hand function. Their basic information was recorded, including basic abilities and pen-holding posture, etc. Using three different angles of 3D printing writing aids, the writing efficiency and the satisfaction of the aids are evaluated by the writing task and the Satisfaction with Assistive Technology.
  Interventions: Behavioral: 3D-printed writing aids task

INTERVENTIONS:
Behavioral: 3D-printed writing aids task — Briefly explain how to wear assistive devices, confirm that the case understands how to operate, and conduct a writing task test. Situation includes no wearable assistive device,three pen placement designs with different angles (5 degrees, 20 degrees, and 30 degrees). Record the writing speed, legibility, posture, and satisfaction of the assistive device after each writing task, etc.

SUMMARY:
Injury to the central or peripheral nerves can lead to limited hand function and further affect the ability of writing. The use of assistive devices can assist writing performance. However, the habit of holding the pen and the ability of the individual case will affect the selection of aids and the efficiency of writing. The 3D printing aids can be individually designed and adjusted to different angles and types. There is no criterion for 3D printing aids decision, often using a case-by-case trial subjective way to confirm, matching takes more time. Aim: To compare the applicability and efficiency of different types of 3D-printed writing aids in nerve injury cases, and to explore which factors affect the choice of aids.

DETAILED DESCRIPTION:
Background: Injury to the central or peripheral nerves can lead to limited hand function and further affect the ability of writing. The use of assistive devices can assist writing performance. However, the habit of holding the pen and the ability of the individual case will affect the selection of aids and the efficiency of writing. The 3D printing aids can be individually designed and adjusted to different angles and types. There is no criterion for 3D printing aids decision, often using a case-by-case trial subjective way to confirm, matching takes more time. Aim: To compare the applicability and efficiency of different types of 3D-printed writing aids in nerve injury cases, and to explore which factors affect the choice of aids.

Methods: Thirty subjects were recruited from outpatient rehabilitation of neurologically injured patients with limited hand function. Their basic information was recorded, including basic abilities, palm and finger size, and pen-holding posture, etc. Using three different angles of 3D printing writing aids, the writing efficiency and the satisfaction of the aids are evaluated by the writing task and the Satisfaction with Assistive Technology. Collected data were analyzed by SPSS (Version 20.0). The significance level of the statistical value is set at 0.05. The basic data and evaluation items of the subjects are observed by descriptive statistical analysis. All the analyzed values will be presented in the form of mean ± standard deviation. The Wilcoxon test is used to compare before and after the use of assistive devices. Data between different aids were analyzed by one-way analysis of variance (ANOVA) with Bonferroni adjustment; basic data and aids choice were analyzed by Pearson's Chi-Square correlation analysis; liner regression was used, and Backward regression was used to confirm whether the variable was removed (p>0.1), and univariate analyses in a general linear manner were used to analyze whether the independent variables of the basic data affected the choice of assistive devices.

ELIGIBILITY:
Inclusion Criteria:

* The medical record shows that the diagnosis is central or peripheral nerve injury, and the onset is more than three months
* The trunk is well controlled and can sit stable on the chair
* The affected hand can control the lifting of the shoulder and the bending of the elbow, and the forearm can be controlled.
* The affected hand is the dominant hand and has difficulty writing

Exclusion Criteria:

* Aged over 75 and under 20
* Cognition or visual perception impairment that affects their ability to copy
* Patients suffer from other diseases of the nervous, cardiopulmonary, and musculoskeletal systems that affect the subject's performance of the movements required by this test.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In cases of central or peripheral nerve injury, symptoms such as sensory paralysis, limited joint mobility, insufficient muscle strength, abnormal tension, unsmooth movements, and lack of segmental movement control may result, affecting the voluntary control of muscles, and showing weak and inaccurate movements. , slowing down, affecting their hand performance, which in turn affects writing tasks
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Writing task | From date of writing task until 4 situations complete, assessed up to 1 session. Each session lasting 60 minutes within one day.
  The individual is asked to copy short sentences in four situations including no wearing aids, writing aids with three angles (5 degrees, 20 degrees, 30 degrees). Calculate the time and quality it takes to complete 10 words. To record its speed, quality (the legibility of the correct number of words, the size of the writing, the number of times it exceeds the line, whether the strength is sufficient and consistent).

SECONDARY OUTCOMES:
Assistive device satisfaction scale | From date of writing task until 4 situations complete, assessed up to 1 session. Each session lasting 60 minutes within one day.
  The questionnaire is a subjective self-filling scale for the use of assistive devices, and the visual analog scale 0-10 scale is used. The items include the writing speed, ease of use, comfort, effectiveness, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Hsinchieh Lee, Master, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armour BS, Courtney-Long EA, Fox MH, Fredine H, Cahill A. Prevalence and Causes of Paralysis-United States, 2013. Am J Public Health. 2016 Oct;106(10):1855-7. doi: 10.2105/AJPH.2016.303270. Epub 2016 Aug 23. PMID 27552260
- [Background] Baronio G, Harran S, Signoroni A. A Critical Analysis of a Hand Orthosis Reverse Engineering and 3D Printing Process. Appl Bionics Biomech. 2016;2016:8347478. doi: 10.1155/2016/8347478. Epub 2016 Aug 9. PMID 27594781
- [Background] Bethoux F. Spasticity Management After Stroke. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):625-39. doi: 10.1016/j.pmr.2015.07.003. Epub 2015 Sep 26. PMID 26522902
- [Background] Chang SH, Chen CL, Yu NY. Biomechanical analyses of prolonged handwriting in subjects with and without perceived discomfort. Hum Mov Sci. 2015 Oct;43:1-8. doi: 10.1016/j.humov.2015.06.008. Epub 2015 Jun 30. PMID 26141665
- [Background] De Stefano, C., Fontanella, F., Impedovo, D., Pirlo, G., & di Freca, A. S. J. P. R. L. (2019). Handwriting analysis to support neurodegenerative diseases diagnosis: A review. 121, 37-45.
- [Background] Hunzeker, M., & Ozelie, R. (2021). A Cost-Effective Analysis of 3D Printing Applications in Occupational Therapy Practice. The Open Journal of Occupational Therapy, 9(1), 1-12.
- [Background] Janson R, Burkhart K, Firchau C, Hicks K, Pittman M, Yopps M, Hatfield S, Garabrant A. Three-dimensional printed assistive devices for addressing occupational performance issues of the hand: A case report. J Hand Ther. 2020 Apr-Jun;33(2):164-169. doi: 10.1016/j.jht.2020.03.025. Epub 2020 May 16. PMID 32423845
- [Background] Jumani, M., Shaikh, S., & Shah, S. A. J. S. I. (2014). RAPID MANUFACTURING TECHNIQUE FOR FABRICATION OF CUSTOM-MADE FOOT ORTHOSES. 26(1).
- [Background] Kuo LC, Hsu HM, Wu PT, Lin SC, Hsu HY, Jou IM. Impact of distal median neuropathy on handwriting performance for patients with carpal tunnel syndrome in office and administrative support occupations. J Occup Rehabil. 2014 Jun;24(2):332-43. doi: 10.1007/s10926-013-9471-8. PMID 23934582
- [Background] Kushki A, Schwellnus H, Ilyas F, Chau T. Changes in kinetics and kinematics of handwriting during a prolonged writing task in children with and without dysgraphia. Res Dev Disabil. 2011 May-Jun;32(3):1058-64. doi: 10.1016/j.ridd.2011.01.026. PMID 21315553
- [Background] Lee KH, Kim DK, Cha YH, Kwon JY, Kim DH, Kim SJ. Personalized assistive device manufactured by 3D modelling and printing techniques. Disabil Rehabil Assist Technol. 2019 Jul;14(5):526-531. doi: 10.1080/17483107.2018.1494217. Epub 2018 Oct 14. PMID 30318956
- [Background] Long TM, Woolverton M, Perry DF, Thomas MJ. Training needs of pediatric occupational therapists in assistive technology. Am J Occup Ther. 2007 May-Jun;61(3):345-54. doi: 10.5014/ajot.61.3.345. PMID 17569392
- [Background] Lubbes, E. (2016). Investigation and Assessment of Upper-Limb Prosthetic Care and Business Model Design for 3D-Printed Prostheses in the Netherlands.
- [Background] Ma HI, Hwang WJ, Tsai PL, Hsu YW. The effect of eating utensil weight on functional arm movement in people with Parkinson's disease: a controlled clinical trial. Clin Rehabil. 2009 Dec;23(12):1086-92. doi: 10.1177/0269215509342334. PMID 19906764
- [Background] Marque P, Gasq D, Castel-Lacanal E, De Boissezon X, Loubinoux I. Post-stroke hemiplegia rehabilitation: evolution of the concepts. Ann Phys Rehabil Med. 2014 Nov;57(8):520-529. doi: 10.1016/j.rehab.2014.08.004. Epub 2014 Aug 23. PMID 25282582
- [Background] Martin, L. M. J. A. J. o. O. T. (1988). Clinical Mechanics of the Hand. 42(3), 199-199.
- [Background] McDonald SS, Levine D, Richards J, Aguilar L. Effectiveness of adaptive silverware on range of motion of the hand. PeerJ. 2016 Feb 15;4:e1667. doi: 10.7717/peerj.1667. eCollection 2016. PMID 26893960
- [Background] Meulenbroek, R. G., & Thomassen, A. J. J. P. R. (1992). Effects of handedness and arm position on stroke-direction preferences in drawing. 54(3), 194-201.
- [Background] Skymne C, Dahlin-Ivanoff S, Claesson L, Eklund K. Getting used to assistive devices: ambivalent experiences by frail elderly persons. Scand J Occup Ther. 2012 Mar;19(2):194-203. doi: 10.3109/11038128.2011.569757. Epub 2011 May 2. PMID 21534712
- [Background] Will, E. J. HANDWRITING, BIOMECHANICS AND SIGNIFICANCE: CONCEPTS IN HANDWRITING IDENTIFICATION.